CLINICAL TRIAL: NCT01074944
Title: A Phase 3, Randomized, Multi-Center, Multi-National, Double-Blind Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Once Daily Versus Twice Daily Dosing of Genz-112638 in Patients With Gaucher Disease Type 1 Who Have Demonstrated Clinical Stability on a Twice Daily Dose of Genz-112638
Brief Title: A Study of Eliglustat Tartrate (Genz-112638) in Patients With Gaucher Disease to Evaluate Once Daily Versus Twice Daily Dosing (EDGE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GZGD03109; 2009-015811-42 (EudraCT Number); EFC12818 (Other: Sanofi)
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Results first posted 2016-12-02 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Gaucher Disease
Keywords: Gaucher disease; Genz-112638; beta-glucosidase; acid β-glucosidase; glucocerebrosidase; glucosylceramide; D-glucosyl-N-acylsphingosine glucohydrolase; substrate reduction therapy
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Twice Daily (BID) Dose Regimen (Experimental): Patients will receive either 50 mg BID or 100 mg BID
  Interventions: Drug: Eliglustat tartrate
- Once Daily (QD) Dose Regimen (Experimental): Patients will receive either 100 mg QD or 200 mg QD
  Interventions: Drug: Eliglustat tartrate

INTERVENTIONS:
Drug: Eliglustat tartrate — Oral Capsule in 50 mg or 100 mg dosages
  Other Names: Genz-112638

SUMMARY:
The primary objective of this study was to evaluate the efficacy and safety of once daily (QD) versus twice daily (BID) dosing of eliglustat tartrate (Genz-112638) in participants with Gaucher disease type 1 who had demonstrated clinical stability on BID dosing of eliglustat tartrate (Genz-112638). The secondary objective was to evaluate the pharmacokinetics (PK) of Genz-99067 when eliglustat tartrate (Genz-112638) was administered QD and BID in participants with Gaucher disease type 1 who had demonstrated clinical stability on BID dosing of eliglustat tartrate (Genz-112638).

DETAILED DESCRIPTION:
NOTE: Other Phase 3 studies being conducted with eliglustat tartrate (Genz-112638) are GZGD02507 (ENGAGE): NCT00891202 and GZGD02607 (ENCORE): NCT00943111

ELIGIBILITY:
Inclusion Criteria:

* The participant who was willing and provided signed informed consent prior to any study-related procedures.
* The participant was ≥18 years of age.
* The participant diagnosed with GD 1 confirmed by a documented deficiency of acid β-glucosidase activity by enzyme assay.
* Female participants of childbearing potential had a documented negative pregnancy test prior to administration of the first dose of eliglustat tartrate (Genz-112638) in this study. In addition, all female participants of childbearing potential used a medically accepted form of contraception throughout the study, i.e., either a barrier method or hormonal contraceptive with norethindrone and ethinyl estradiol or similar active components
* The participant met all of the following criteria at the time of screening: hemoglobin level ≥9 g/dL (mean of 2 measurements); platelet count ≥70,000/mm^3 (mean of 2 measurements); spleen volume ≤25 multiples of normal (MN); liver volume ≤2.0 MN.
* The participant consented to provide a blood sample for genotyping for Gaucher disease and for CYP2D6 to categorize the participant's predicted rate of metabolism, if these genotyping results were not already available for the participant.
* The participant was willing to abstain from consumption of grapefruit, grapefruit juice, or grapefruit products for 72 hours prior to administration of the first dose of Genz-112638 and throughout the duration of the study.

Exclusion Criteria:

* The participant was participating in GZGD02607 study, "A Phase 3, Randomized, Multi-Center, Multi-National, Open-Label, Active Comparator Study to Evaluate the Efficacy and Safety of Genz-112638 in Participants with GD1 who have been Stabilized with Cerezyme ® ," or was eligible for inclusion in GZGD02607 (while enrollment was ongoing) and had access to a physician participating in GZGD02607, or the participant was participating in GZGD02507 study, "A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study Confirming the Efficacy and Safety of Genz-112638 in Participants with GD1," or was eligible for inclusion in GZGD02507 (while enrollment was ongoing) and had access to a physician participating in GZGD02507.
* The participant received miglustat within 6 months prior to administration of the first dose of Genz-112638 in this study.
* The participant had a partial or total splenectomy within 3 years prior to randomization.
* The participant received pharmacological chaperones or miglustat within 6 months prior to administration of the first dose of eliglustat tartrate (Genz-112638) in this study.
* The participant had any evidence of neurologic disorder (e.g., peripheral neuropathy, tremor, seizures, Parkinsonism or cognitive impairment) or pulmonary involvement (e.g., pulmonary hypertension) as related to Gaucher disease.
* The participant was transfusion-dependent.
* The participant had a documented deficiency of iron, vitamin B-12, or folate that requires treatment not yet initiated or, if initiated, the participant had not been stable under treatment for at least 3 months prior to administration of the first dose of Genz-112638 in this study.
* The participant had documented prior esophageal varices or clinically significant liver infarction or current liver enzymes (alanine transaminase [ALT]/aspartate aminotransferase [AST]) or total bilirubin >2 times the upper limit of normal (ULN), unless the participant had a diagnosis of Gilbert Syndrome.
* The participant had any clinically significant disease, other than Gaucher disease, including cardiovascular, renal, hepatic, gastrointestinal, pulmonary, neurologic, endocrine, metabolic (including hypokalaemia or hypomagnesemia), or psychiatric disease, other medical conditions, or serious intercurrent illnesses that, in the opinion of the Investigator, precluded participation in the study.
* The participant was known to have any of the following: Clinically significant coronary artery disease including history of myocardial infarction [MI] or ongoing signs or symptoms consistent with cardiac ischemia or heart failure; or clinically significant arrhythmias or conduction defect such as 2nd or 3rd degree AV block, complete bundle branch block, prolonged QTc interval, or sustained ventricular tachycardia (VT).
* The participant who tested positive for the human immunodeficiency virus (HIV) antibody, Hepatitis C antibody, or Hepatitis B surface antigen.
* The participant received an investigational product (other than eliglustat tartrate (Genz-112638)) within 30 days prior to administration of the first dose of eliglustat tartrate (Genz-112638) in this study.
* The participant was scheduled for in-participant hospitalization, including elective surgery, during the study.
* The participant had a history of cancer, with the exception of basal cell carcinoma, within 5 years prior to administration of the first dose of Genz-112638 in this study.
* The participant was pregnant or lactating.
* The participant had received any medication that may cause QTc interval prolongation within 30 days prior to the first dose of Genz-112638. Exception: Diphenhydramine (Benadryl) or other medications used as premedication for ERT infusions were allowed up to 7 days prior to the first dose of Genz-112638.
* The participant had received for the first time (i.e., the participant was not already chronically using) any of the following medications within 30 days prior to the first dose of Genz-112638:

  * Strong inhibitors of CYP2D6 or CYP3A4;
  * Inducers of CYP3A4. Exception: Premedications for ERT infusions were allowed up to 7 days prior to the first dose of Genz-112638.
* The participant was a CYP2D6 non-poor metabolizer or an indeterminate metabolizer with one allele identified as active who was chronically receiving both a strong competitive inhibitor of CYP2D6 and a strong competitive inhibitor of CYP3A4 and for whom no reasonable alternative medication exists. or
* The participant was a CYP2D6 poor metabolizer or an indeterminate metabolizer with neither allele known to be active who was chronically receiving a strong competitive inhibitor of CYP3A4 and for whom no reasonable alternative medication exists.

Exception for both cases: Premedications for ERT infusions were allowed up to 7 days prior to the first dose of Genz-112638.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (46):
- United States (10):
  - University of California, San Diego Medical Center, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University Medical Center, Decatur, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Mount Sinai Medical Center, New York, New York
  - New York University School of Medicine, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - O and O Alpan LLC, Springfield, Virginia
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown
  - Monash Medical Centre, Clayton, VIC
  - Royal Perth Hospital, Perth, WA
- Medical University Vienna, Vienna, Austria
- Brazil (9):
  - Hospital das Clinicas da UFMG, Belo Horizonte
  - Cettro - Centro de Tratamento de Oncologia e Hematologia, Brasília
  - Hemocentro - UNICAMP, Campinas
  - Instituto Tropical de Medicina Reprodutiva e Menopausa - INTRO, Cuiabá
  - Hospital Universitario Walter Cantidio - HUWC, Fortaleza
  - Hemocentro de Ribeirão Preto Núcleo de Hemoterapia de Franca, Franca
  - Hemorio, Rio de Janeiro
  - Hospital de Clínicas da Universidade Federal do Parana, São Paulo
  - IGEIM - Institute of Genetic and Inborn Erros of Metabolism, São Paulo
- Mount Sinai Hospital, Toronto, Canada
- China (4):
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Shanghai Xinhua Hospital Shanghai Xinhua Hospital, Shanghai
  - Tianjin Hematonosis Hospital, Tianjin
- University Hospital Centre Zagreb, Zagreb, Croatia
- France (2):
  - Hôpital Haut Lévêque, Bordeaux
  - Hôpital Femme Mère Enfant Centre de référence des maladies Héréditaires du métabolisme, Bron
- General Hospital of Athens "G. Gennimatas", Athens, Greece
- King Edward Memorial (KEM) Hospital, Mumbai, India
- Japan (4):
  - Hiroshima University Hospital, Hiroshima
  - Jikei University Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Mie Chuou Medical Center, Tsu, Mie
- Academic Medical Center, Amsterdam, Netherlands
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Hospital do Divíno Espírito Santo, Ponta Delgada - São Miguel - Açores
- Spitaulu Clinic de Urgenta, Cluj-Napoca, Romania
- Russia (3):
  - State Medical and Prophylactic Healthcare Institution; Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - Hematology Research Center of Russian Academy of Medical Sciences, Moscow
  - St. Petersburg State Medical Pavlov University, Saint Petersburg
- Clinical Centre of Serbia, Belgrade, Serbia
- University Hospital Lund, Lund, Sweden

REFERENCES:
- [Background] McEachern KA, Fung J, Komarnitsky S, Siegel CS, Chuang WL, Hutto E, Shayman JA, Grabowski GA, Aerts JM, Cheng SH, Copeland DP, Marshall J. A specific and potent inhibitor of glucosylceramide synthase for substrate inhibition therapy of Gaucher disease. Mol Genet Metab. 2007 Jul;91(3):259-67. doi: 10.1016/j.ymgme.2007.04.001. Epub 2007 May 16. PMID 17509920
- [Background] Lukina E, Watman N, Arreguin EA, Banikazemi M, Dragosky M, Iastrebner M, Rosenbaum H, Phillips M, Pastores GM, Rosenthal DI, Kaper M, Singh T, Puga AC, Bonate PL, Peterschmitt MJ. A phase 2 study of eliglustat tartrate (Genz-112638), an oral substrate reduction therapy for Gaucher disease type 1. Blood. 2010 Aug 12;116(6):893-9. doi: 10.1182/blood-2010-03-273151. Epub 2010 May 3. PMID 20439622
- [Background] Lukina E, Watman N, Arreguin EA, Dragosky M, Iastrebner M, Rosenbaum H, Phillips M, Pastores GM, Kamath RS, Rosenthal DI, Kaper M, Singh T, Puga AC, Peterschmitt MJ. Improvement in hematological, visceral, and skeletal manifestations of Gaucher disease type 1 with oral eliglustat tartrate (Genz-112638) treatment: 2-year results of a phase 2 study. Blood. 2010 Nov 18;116(20):4095-8. doi: 10.1182/blood-2010-06-293902. Epub 2010 Aug 16. PMID 20713962
- [Derived] Charrow J, Fraga C, Gu X, Ida H, Longo N, Lukina E, Nonino A, Gaemers SJM, Jouvin MH, Li J, Wu Y, Xue Y, Peterschmitt MJ. Once- versus twice-daily dosing of eliglustat in adults with Gaucher disease type 1: The Phase 3, randomized, double-blind EDGE trial. Mol Genet Metab. 2018 Mar;123(3):347-356. doi: 10.1016/j.ymgme.2017.12.001. Epub 2018 Jan 4. PMID 29358012
- See also: GZGD02507 (NCT00891202) eliglustat tartrate (Genz-112638) Phase 3 Clinical Study in untreated patients with Gaucher disease type 1 — http://clinicaltrials.gov/ct2/show/NCT00891202?term=genz+ENGAGE&rank=1
- See also: GZGD02607 (NCT00943111) eliglustat tartrate (Genz-112638) Phase 3 Clinical Study in patients with Gaucher disease type 1 who have been stabilized on Cerezyme — http://clinicaltrials.gov/ct2/show/NCT00943111?term=genz+encore&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 45 centers in 17 countries between 1 June 2010 and 6 October 2015. A total of 219 participants were screened, out of which 170 entered into the lead in period (LIP). Remaining 48 participants were screen failures and 1 participant withdrew before entering into the LIP.
Pre-assignment Details: Participant flow divided into 4 periods: LIP:to assess randomization criteria. Primary analysis period (PAP):to assess therapeutic efficacy at 2 dosing regimen in randomized participants. Long-term treatment period (LTTP): to assess long term efficacy. Extended treatment period (ETP):those who were non-randomized after LIP continued in this period.
Groups:
- LIP, Eliglustat: All participants (except in Japan) received eliglustat 50 mg, twice daily (BID) on Day 1 titrated up to 100 mg BID (50 or 100 mg capsules) based on their individual pharmacokinetics (PK) data for up to 78 weeks. All participants in Japan received eliglustat 50 mg once only on Day 1 and then eliglustat 50 mg BID from Day 2 titrated up to 100 mg BID (50 or 100 mg capsules) based on their individual PK data for up to 78 weeks.
- PAP, Eliglustat: Once Daily: All participants who were randomized after meeting all randomization criteria (defined as: no more than 1 bone crisis and was free of other clinically symptomatic bone disease [such as bone pain attributable to osteonecrosis and/or pathological fractures) during the first 6 months of the LIP; mean hemoglobin level of ≥11 g/dL [if female] and ≥12 g/dL [if male]; mean platelet count ≥100,000/mm^3; spleen volume ≤10 times of normal; liver volume ≤1.5 times of normal; had a dose of 50 mg BID or 100 mg BID of eliglustat for at least 4 months and a peak (2-hour) Genz-99067 plasma concentration of <50 ng/mL) after either 26, 52 or 78 weeks of LIP received eliglustat capsules at the total daily dose (TDD) of 100 mg or 200 mg (the TDD they were on before randomization) once daily (QD) from Day 1 up to Week 52 in PAP (50 or 100 mg capsules).
- PAP, Eliglustat: Twice Daily: All participants who were randomized after meeting all randomization criteria (defined as: no more than 1 bone crisis and was free of other clinically symptomatic bone disease [such as bone pain attributable to osteonecrosis and/or pathological fractures) during the first 6 months of the LIP; mean hemoglobin level of ≥11 g/dL [if female] and ≥12 g/dL [if male]; mean platelet count ≥100,000/mm^3; spleen volume ≤10 times of normal; liver volume ≤1.5 times of normal; had a dose of 50 mg BID or 100 mg BID of eliglustat for at least 4 months and a peak (2-hour) Genz-99067 plasma concentration of <50 ng/mL) after either 26, 52 or 78 weeks of LIP, received eliglustat at the TDD 50 mg BID or 100 mg BID (the TDD they were on before randomization) from Day 1 up to Week 52 in PAP (50 or 100 mg capsules).
- LTTP, Eliglustat: All participants who entered PAP continued their blinded randomized treatment for first 4 weeks. Participants who at Week 52 of PAP maintained their therapeutic goals (defined as: no more than 2 bone crisis during PAP [with no more than 1 bone crisis during either first 6 months or later 6 months of PAP] and is free of other clinically symptomatic bone disease during PAP; hemoglobin level not decreased by >1.5 g/dL from Baseline for PAP [defined as last available assessment prior to randomization]; platelet count not decreased by >25% from Baseline for PAP; spleen volume not increased by 25% from Baseline for PAP; liver volume not increased by >20% from Baseline for PAP), continued into the LTTP and received their TDD of eliglustat (100 mg or 200 mg) QD till the end of the study. The participants who did not maintain all their therapeutic goals continued into the LTTP and received their TDD of eliglustat (100 mg or 200 mg) BID till the end of the study.
- ETP, Eliglustat: All participants who did not meet all the randomization criteria at Week 78 of the LIP continued in the ETP and received eliglustat capsules at the same dose as they were receiving at the end of LIP till the end of the study.
Period: Lead-in Period (up to 78 Weeks)
Arm/Group | LIP, Eliglustat | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily | LTTP, Eliglustat | ETP, Eliglustat
Started | 170 (LIP conducted to assess randomization criteria of all participants in single reporting arm.) | 0 | 0 | 0 | 0
Completed | 157 | 0 | 0 | 0 | 0
Not Completed | 13 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0
Not completed — Non-Compliance With Protocol | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0 | 0 | 0
Period: Primary Analysis Period (up to 52 Weeks)
Arm/Group | LIP, Eliglustat | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily | LTTP, Eliglustat | ETP, Eliglustat
Started | 0 | 65 (Participants who were randomized after LIP received treatment in PAP.) | 66 (Participants who were randomized after LIP received treatment in PAP.) | 0 | 0
Completed | 0 | 54 | 60 | 0 | 0
Not Completed | 0 | 11 | 6 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 3 | 0 | 0
Not completed — Treatment Failure | 0 | 6 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0
Not completed — Non-Compliant to Protocol | 0 | 1 | 1 | 0 | 0
Period: Long Term Treatment
Arm/Group | LIP, Eliglustat | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily | LTTP, Eliglustat | ETP, Eliglustat
Started | 0 | 0 | 0 | 121 (Participants who completed PAP (114) including those who considered as treatment failure in PAP (7).) | 0
Completed | 0 | 0 | 0 | 95 | 0
Not Completed | 0 | 0 | 0 | 26 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0
Not completed — Transitioned to Commercial Eliglustat | 0 | 0 | 0 | 18 | 0
Not completed — Entered in Period, But Not Treated | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0
Period: Extended Treatment (up to 42 Months)
Arm/Group | LIP, Eliglustat | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily | LTTP, Eliglustat | ETP, Eliglustat
Started | 0 | 0 | 0 | 0 | 25 (Participants who were failed to meet the randomization criteria during the lead-in period.)
Completed | 0 | 0 | 0 | 0 | 20
Not Completed | 0 | 0 | 0 | 0 | 5
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 2
Not completed — Transitioned to Commercial Eliglustat | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: All treated (AT) analysis set included all participants who received at least 1 dose of eliglustat during LIP.
Groups:
- All Participants: All participants who received treatment in LIP (eliglustat 50 mg BID on Day 1 titrated up to 100 mg BID [50 or 100 mg capsules] based on their individual PK data for up to 78 weeks [except for the participants in Japan]. Participants in Japan received eliglustat 50 mg once only on Day 1 and then eliglustat 50 mg BID from Day 2 titrated up to 100 mg BID [50 or 100 mg capsules] based on their individual PK data for up to 78 weeks) and assessed for randomization.
Arm/Group | All Participants
Number analyzed (Participants) | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (15.1)
Gender [Count of Participants; unit: Participants]
  Female | 81
  Male | 89

OUTCOME MEASURES:

1. Primary Outcome: PAP: Percentage of Participants Who Remained Stable for 52 Weeks During the PAP
Description: Participants were considered as stable if they met all of the following criteria: 1) no more than 2 bone crisis during PAP (with no more than 1 bone crisis during either the first 6 months or the later 6 months of the period), and were free of other clinically symptomatic bone disease during the entire 52-week PAP; 2) hemoglobin level not decreased >1.5 g/dL from Baseline for PAP; 3) platelet count not decreased >25% from Baseline for PAP; 4) spleen volume (in multiples of normal [MN]) did not increase >25% from Baseline for PAP; 5) liver volume (in MN) did not increase >20% from Baseline for PAP. Baseline for PAP was defined as the last assessment prior to randomization.
Time Frame: PAP Baseline up to the end of PAP (Week 52)
Population: Analysis was performed on per protocol (PP) population which included all participants who were at least 80% compliant with investigational medicinal product (IMP) dosing during PAP, had all of the necessary Baseline and Week 52 assessments to evaluate the primary endpoint, and did not have major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PAP, Eliglustat: Once Daily: All participants who were randomized after either 26, 52 or 78 weeks of LIP received eliglustat at the TDD of 100 mg or 200 mg (the TDD they were on before randomization) QD from Day 1 up to Week 52 in PAP (50 or 100 mg capsules).
- PAP, Eliglustat: Twice Daily: All participants who were randomized after either 26, 52 or 78 weeks of LIP received eliglustat 50 mg BID or 100 mg BID (the TDD they were on before randomization) from Day 1 up to Week 52 in PAP (50 or 100 mg capsules).
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
percentage of participants | 80.4 [67.6 to 89.8] | 83.1 [71.0 to 91.6]
Statistical Analysis 1: Comparison: PAP, Eliglustat: Once Daily vs PAP, Eliglustat: Twice Daily; Test type: Non-Inferiority or Equivalence — Eliglustat QD treatment was declared non-inferior to BID treatment if the lower bound of the 95% confidence interval (CI) for the difference was within the non-inferiority margin of -0.15 (or -15%); Difference in Percentage Stable = -2.7, 95% CI 2-sided [-17.7 to 11.9]

2. Secondary Outcome: PAP: Mean Hemoglobin (Hb) Level at Baseline, Weeks 26 and 52
Time Frame: Baseline, Week 26, Week 52
Population: PP population included all participants who were at least 80% compliant with IMP dosing during PAP, had all of the necessary Baseline and Week 52 assessments to evaluate the primary endpoint, and did not have major protocol deviations. Here 'n' signifies number of participants with available data at specified time points for each arm respectively.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
g/dL
  Baseline (n=56, 59) | 13.641 (1.214) | 13.691 (1.273)
  Week 26 (n=56, 57) | 13.677 (1.377) | 13.946 (1.509)
  Week 52 (n=56, 59) | 13.605 (1.432) | 13.824 (1.442)

3. Secondary Outcome: PAP: Mean Platelet Count at Baseline, Weeks 26, 52
Time Frame: Baseline, Week 26, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: platelets*10^9 /L
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
platelets*10^9 /L
  Baseline (n=56, 59) | 204.01 (81.49) | 171.09 (63.50)
  Week 26 (n=56, 57) | 195.75 (66.65) | 173.94 (65.61)
  Week 52 (n=56, 59) | 207.20 (80.62) | 176.10 (62.01)

4. Secondary Outcome: PAP: Mean Spleen Volume at Baseline, Weeks 26, 52
Time Frame: Baseline, Week 26, Week 52
Population: PP population included all participants who were at least 80% compliant with IMP dosing during PAP, had all of the necessary Baseline and Week 52 assessments to evaluate the primary endpoint, and did not have major protocol deviations. Here 'n' signifies number of participants with available data for specified category for each arm respectively.
Measure: Mean (Standard Deviation); unit: MN
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
MN
  Baseline (n= 39, 45) | 3.309 (1.465) | 3.787 (1.623)
  Week 26 (n= 39, 45) | 3.066 (1.299) | 3.504 (1.365)
  Week 52 (n= 39, 45) | 3.017 (1.381) | 3.394 (1.305)

5. Secondary Outcome: PAP: Mean Liver Volume at Baseline, Weeks 26, 52
Time Frame: Baseline, Week 26 and Week 52
Population: PP population included all participants who were at least 80% compliant with IMP dosing during PAP, had all of the necessary Baseline and Week 52 assessments to evaluate the primary endpoint, and did not have major protocol deviations.
Measure: Mean (Standard Deviation); unit: MN
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
MN
  Baseline (n=56, 59) | 0.981 (0.187) | 1.040 (0.198)
  Week 26 (n=56, 59) | 0.987 (0.190) | 1.024 (0.179)
  Week 52 (n=56, 59) | 0.970 (0.170) | 1.009 (0.196)

6. Secondary Outcome: PAP: Mean Biomarker (Chitotriosidase) Value at Baseline, Weeks 26 and Week 52
Description: Chitotriosidase biomarker was assayed from plasma.
Time Frame: Baseline, Week 26, Week 52
Population: PP population which all participants who were at least 80% compliant with IMP dosing during PAP, had all of the necessary Baseline and Week 52 assessments to evaluate the primary endpoint, and did not have major protocol deviations. Here, 'n' signifies number of participants with available data for specified category for each arm respectively.
Measure: Mean (Standard Deviation); unit: nmol/hr/mL
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
nmol/hr/mL
  Baseline (n=55, 59) | 1523.7 (2556.6) | 1554.9 (1895.0)
  Week 26 (n=52, 54) | 1279.6 (2328.1) | 1242.0 (2012.6)
  Week 52 (n=54, 55) | 1076.6 (1855.8) | 1170.1 (1683.3)

7. Secondary Outcome: PAP: Mean Biomarker (GL-1 on DBS) Value at Baseline, Week 26 and Week 52
Description: GL-1 on DBS biomarker was assayed from dried blood spot (DBS).
Time Frame: Baseline, Week 26 and week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
mcg/mL
  GL-1 on DBS: Baseline (n=54, 55) | 2.257 (0.835) | 2.425 (1.378)
  GL-1 on DBS: week 26 (n=54, 54) | 2.481 (1.037) | 2.563 (1.100)
  GL-1 on DBS: week 52 (n=53, 55) | 2.853 (1.383) | 2.707 (1.443)

8. Secondary Outcome: PAP: Mean Biomarker Macrophage Inflammatory Protein-1 Beta (MIP1-beta) Value at Baseline, Weeks 26, 52
Description: MIP1-beta biomarker was assayed from plasma.
Time Frame: Baseline, Week 26, Week 52
Population: PP population included all participants who were at least 80% compliant with dosing during PAP, had all of the necessary Baseline and Week 52 assessments to evaluate the primary endpoint, and did not have major protocol deviations. Here, 'n' signifies number of participants with available data for specified category for each arm respectively.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
pg/mL
  Baseline (n=54, 58) | 77.7 (74.4) | 118.8 (156.3)
  Week 26 (n=52, 54) | 74.5 (68.0) | 121.0 (204.4)
  Week 52 (n=54, 55) | 81.3 (82.8) | 117.9 (165.3)

9. Secondary Outcome: PAP: Bone Mineral Density (BMD) at Baseline and Week 52
Description: BMD measurements of the spine and bilateral femur were acquired by dual-energy x-ray absorptiometry (DXA) scan.
Time Frame: Baseline, Week 52
Population: PP population included all participants who were at least 80% compliant with IMP dosing during PAP, had all of the necessary Baseline and Week 52 assessments to evaluate the primary endpoint, and did not have major protocol deviations. Here, 'n' signifies number of participants with available data at specified time points for each arm respectively.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
g/cm^2
  Lumbar Spine: Baseline (n=51, 55) | 1.073 (0.177) | 1.081 (0.172)
  Lumbar Spine: Week 52 (n=51, 55) | 1.089 (0.183) | 1.086 (0.177)
  Left Femur: Baseline (n=48, 47) | 0.979 (0.219) | 1.000 (0.199)
  Left Femur: Week 52 (n=48, 47) | 0.972 (0.211) | 0.990 (0.196)
  Right Femur: Baseline (n=48, 47) | 0.971 (0.217) | 0.996 (0.184)
  Right Femur: Week 52 (n=48, 47) | 0.967 (0.213) | 0.981 (0.177)

10. Secondary Outcome: PAP: Total T-Scores for BMD at Baseline and Week 52
Description: Images of the spine and bilateral femur were obtained by DXA to determine T-score for each bone area and total bone mineral density. The T-score bone density categories were: normal (score >-1), osteopenia (score -2.5 to <=-1), and osteoporosis (score <= -2.5).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
T-score
  Lumbar Spine T-Score: Baseline (n=49, 52) | -0.722 (1.415) | -0.771 (1.217)
  Lumbar Spine T-Score: Week 52 (n=49, 52) | -0.580 (1.476) | -0.717 (1.271)
  Left Femur T-Score: Baseline (n=46, 44) | -0.459 (1.385) | -0.368 (1.347)
  Left Femur T-Score: Week 52 (n=46, 44) | -0.509 (1.342) | -0.441 (1.326)
  Right Femur T-score: Baseline (n=46, 44) | -0.574 (1.327) | -0.382 (1.282)
  Right Femur T-score: Week 52 (n=46, 44) | -0.607 (1.308) | -0.530 (1.236)

11. Secondary Outcome: PAP: Total Z-scores for BMD at Baseline and Week 52
Description: Images of the spine and bilateral femur were obtained by DXA to determine Z-score for each bone area and total bone mineral density. The Z-score bone density categories are: normal (score >-2) and below normal (score <=-2).
Time Frame: Baseline, Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
Z-score
  Lumbar Spine Z-scores: Baseline (n=51, 55) | -0.492 (1.517) | -0.609 (1.166)
  Lumbar Spine Z-scores: Week 52 (n=51, 55) | -0.324 (1.559) | -0.555 (1.202)
  Left Femur Z-scores: Baseline (n= 48, 47) | -0.171 (1.316) | -0.115 (1.294)
  Left Femur Z-scores: Week 52 (n= 48, 47) | -0.202 (1.250) | -0.183 (1.274)
  Right Femur Z-scores: Baseline (n= 48, 47) | -0.235 (1.251) | -0.140 (1.194)
  Right Femur Z-scores: Week 52 (n= 48, 47) | -0.248 (1.214) | -0.260 (1.141)

12. Secondary Outcome: PAP: Number of Participants With Mobility Status Asessments (MS) at Baseline, Weeks 26, and 52.
Description: Mobility, i.e., ability to walk was assessed as a part of Gaucher disease assessment in participants. In this outcome, number of participants with their different mobility status along with the use of mobility aids (unrestricted mobility, walks with difficulty, walks with orthopaedic aid, requires wheelchair, bedridden) at specified time points were reported.
Time Frame: Baseline, Week 26 and Week 52
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
participants
  MS, Unrestricted: Baseline (n=56, 59) | 49 | 59
  MS, Unrestricted: Week 26 (n=55, 57) | 46 | 56
  MS, Unrestricted: Week 52 (n=51, 58) | 50 | 57
  MS, Walks with Difficulty: Baseline (n=56, 59) | 6 | 0
  MS, Walks with Difficulty: Week 26 (n=55, 57) | 8 | 1
  Ms, Walks with Difficulty: Week 52 (n=51, 58) | 5 | 1
  MS, Walks with Orthopedic Aid: Baseline (n=56, 59) | 1 | 0
  MS, Walks with Orthopedic Aid: Week 26 (n=55, 57) | 1 | 0
  MS, Walks with Orthopedic Aid: Week 52 (n=51, 58) | 0 | 0
  MS, Required Wheelchair: Baseline (n=56, 59) | 0 | 0
  MS, Required Wheelchair: Week 26 (n=55, 57) | 0 | 0
  MS, Required Wheelchair: Week 52 (n=51, 58) | 1 | 0
  MS, Bedridden: Baseline (n=56, 59) | 0 | 0
  MS, Bedridden: Week 26 (n=55, 57) | 0 | 0
  MS, Bedridden: Week 52 (n=51, 58) | 0 | 0

13. Secondary Outcome: PAP: Number of Participants With Bone Crises at Baseline, Weeks 26 and 52
Description: Bone crisis was assessed as a part of Gaucher disease assessment in participants. Acute, excruciating episodic bone pain is characteristic of Gaucher bone crisis, which typically causes debilitation lasting several days or longer and requires treatment with immobilization, hydration, and opioid analgesics. Participants were categorized as 0= no bone crisis, 1= 1 bone crisis, and 2= 2 bone crises during the assessment period. In this outcome, number of participants with different bone crises levels at specified time points were reported.
Time Frame: Baseline, Week 26, and Week 52
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
participants
  Bone Crisis (0): Baseline (n=56, 59) | 55 | 57
  Bone Crisis (0): Week 26 (n=55,57) | 54 | 56
  Bone Crisis (0): Week 52 (n=56, 58) | 56 | 57
  Bone Crisis (1): Baseline (n=56, 59) | 1 | 2
  Bone Crisis (1): Week 26 (n=55, 57) | 0 | 1
  Bone Crisis (1): Week 52 (n=56, 58) | 0 | 1
  Bone Crisis (2): Baseline (n=56, 59) | 0 | 0
  Bone Crisis (2): week 26 (n=55, 57) | 1 | 0
  Bone Crisis (2): week 52 (n=56, 58) | 0 | 0

14. Secondary Outcome: PAP: Number of Participants With Bone Pain Levels During the Past 4 Weeks at Baseline, Weeks 26 and 52
Description: Bone pain was assessed as a part of Gaucher disease assessment in participants. Participants were categorized as none (no bone pain), very mild bone pain, mild bone pain, moderate bone pain, severe bone pain and extreme bone pain during the past 4 weeks. In this outcome, number of participants with different level of bone pain during the past 4 weeks at specified time points were reported.
Time Frame: Baseline, Week 26, and Week 52
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
participants
  None: Baseline (n=56, 59) | 42 | 49
  None: Week 26 (n=55, 57) | 42 | 49
  None: Week 52 (n=56, 58) | 41 | 45
  Very Mild: Baseline (n=56, 59) | 2 | 1
  Very Mild: Week 26 (n=55, 57) | 3 | 4
  Very Mild: Week 52 (n=56, 58) | 3 | 7
  Mild: Baseline (n=56, 59) | 7 | 3
  Mild: Week 26 (n=55, 57) | 5 | 3
  Mild: Week 52 (n=56, 58) | 6 | 2
  Moderate: Baseline (n=56, 59) | 4 | 5
  Moderate: Week 26 (n=55, 57) | 5 | 1
  Moderate: Week 52 (56, 58) | 6 | 2
  Severe: Baseline (n=56, 59) | 1 | 1
  Severe: Week 26 (n=55, 57) | 0 | 0
  Severe: Week 52 (n=56, 58) | 0 | 2
  Extreme: Baseline (n=56, 59) | 0 | 0
  Extreme: Week 26 (n=55, 57) | 0 | 0
  Extreme: Week 52 (n=56, 58) | 0 | 0

15. Secondary Outcome: PAP: Total Bone Marrow Burden Score (BMB) at Baseline and Week 52
Description: BMB Score was measured using magnetic resonance imaging (MRI), range from 0 (no abnormalities) to 8 points (severe disease) for the lumbar spine and from 0 (no abnormalities) to 8 points (severe disease) for the femurs. The total score was calculated as the sum of scores for femur and lumbar spine regions which ranged from 0 (no abnormalities) -16 (severe disease) points. A higher BMB score signified more severe bone marrow involvement.
Time Frame: Baseline, Week 52
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: BMB Score
Arm/Group | PAP, Eliglustat: Once Daily | PAP, Eliglustat: Twice Daily
Number analyzed (Participants) | 56 | 59
BMB Score
  BMB Score: Baseline (n=52, 49) | 8.276 (2.891) | 9.136 (2.784)
  BMB Score: Week 52 (n=51, 48) | 7.971 (2.689) | 8.705 (2.633)

16. Secondary Outcome: LIP: Mean Hemoglobin (Hb) Level at Baseline, Weeks 26, 52 and 78
Time Frame: Baseline, Week 26, Week, 52, and Week 78
Population: Analysis was performed on all treated (AT) analysis set which included all participants who received at least 1 dose of eliglustat during lead in period. Here 'n' signifies number of participants with available data at specified time points.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- LIP: Eliglustat: All participants (except in Japan) received eliglustat 50 mg BID on Day 1 titrated up to 100 mg BID (50 or 100 mg capsules) based on their individual PK data for up to 78 weeks. All participants in Japan received eliglustat 50 mg once only on Day 1 and then eliglustat 50 mg BID from Day 2 titrated up to 100 mg BID (50 or 100 mg capsules) based on their individual PK data for up to 78 weeks.
Arm/Group | LIP: Eliglustat
Number analyzed (Participants) | 170
g/dL
  Baseline (n=170) | 13.435 (1.560)
  Week 26 (n=163) | 13.443 (1.382)
  Week 52 (n=74) | 13.434 (1.497)
  Week 78 (n=41) | 13.329 (1.528)

17. Secondary Outcome: LIP: Mean Platelet Count at Baseline, Weeks 26, 52 and 78
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: Analysis was performed on AT analysis set which included all participants who received at least 1 dose of eliglustat during LIP. Here 'n' signifies number of participants with available data at specified time points.
Measure: Mean (Standard Deviation); unit: platelets*10^9 /L
Arm/Group | LIP: Eliglustat
Number analyzed (Participants) | 170
platelets*10^9 /L
  Baseline (n=170) | 178.653 (92.732)
  Week 26 (n=163) | 180.021 (85.426)
  Week 52 (n=74) | 176.378 (79.880)
  Week 78 (n=41) | 168.720 (74.117)

18. Secondary Outcome: LIP: Mean Liver Volume at Baseline, Weeks 26, 52 and 78
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: Analysis was performed on AT participants which included all participants who received at least 1 dose of eliglustat during lead in period. Here, 'n' signifies number of participants with available data at specified time points.
Measure: Mean (Standard Deviation); unit: MN
Arm/Group | LIP: Eliglustat
Number analyzed (Participants) | 170
MN
  Baseline (n=170) | 1.044 (0.243)
  Week 26 (n=149) | 1.040 (0.229)
  Week 52 (n=68) | 1.059 (0.242)
  Week 78 (n=39) | 1.062 (0.236)

19. Secondary Outcome: LIP: Mean Spleen Volume at Baseline, Weeks 26, 52 and 78
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: Analysis was performed on AT participants which included all participants who received at least 1 dose of eliglustat during lead in period. Here 'n' signifies number of participants with available data at specified time points.
Measure: Mean (Standard Deviation); unit: MN
Arm/Group | LIP: Eliglustat
Number analyzed (Participants) | 170
MN
  Baseline (n=119) | 4.448 (2.314)
  Week 26 (n=106) | 3.840 (1.801)
  Week 52 (n=52) | 4.094 (1.767)
  Week 78 (n=30) | 4.088 (2.089)

20. Secondary Outcome: LIP: Mean Biomarker (Chitotriosidase) Value at Baseline, Weeks 26, 52, and 78
Description: Chitotriosidase biomarker was assayed from plasma.
Time Frame: Baseline, Week 26, Week 52 and Week 78
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nmol/hr/mL
Groups:
- LIP: Eliglustat: All participants (except in Japan) received eliglustat 50 mg, twice daily (BID) on Day 1 titrated up to 100 mg BID (50 or 100 mg capsules) based on their individual PK data for up to 78 weeks. All participants in Japan received eliglustat 50 mg once only on Day 1 and then eliglustat 50 mg BID from Day 2 titrated up to 100 mg BID (50 or 100 mg capsules) based on their individual PK data for up to 78 weeks.
Arm/Group | LIP: Eliglustat
Number analyzed (Participants) | 170
nmol/hr/mL
  Chitotriosidase: Baseline (n=170) | 2437.92 (3291.25)
  Chitotriosidase: week 26 (n=157) | 1802.93 (2529.29)
  Chitotriosidase: week 52 (n=72) | 1755.70 (2649.14)
  Chitotriosidase: week 78 (n=41) | 1677.02 (2718.75)

21. Secondary Outcome: LIP: Mean Biomarker (GL-1 on DBS) Value at Baseline, Week 26, Week 52, and Week 78
Description: GL-1 on DBS biomarker was assayed from dried blood spot.
Time Frame: Baseline, Week 26, Week 52 and Week 78
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | LIP: Eliglustat
Number analyzed (Participants) | 170
mcg/mL
  GL-1 on DBS: Baseline (n=159) | 4.358 (2.155)
  GL-1 on DBS: Week 26 (n=144) | 2.340 (0.868)
  GL-1 on DBS: Week 52 (n=68) | 2.279 (0.730)
  GL-1 on DBS: Week 78 (n=39) | 2.495 (1.500)

22. Secondary Outcome: LIP: Mean Biomarker (MIP1-beta) Value at Baseline, Week 78
Description: MIP1-beta biomarker was assayed from plasma.
Time Frame: Baseline and Week 78
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LIP: Eliglustat
Number analyzed (Participants) | 170
pg/mL
  MIP-1beta: Baseline (n=170) | 142.433 (125.961)
  MIP-1beta: Week 78 (n=41) | 132.180 (189.454)

23. Secondary Outcome: LIP: Number of Participants With Mobility Status (MS) at Baseline, Weeks 26, 52 and 78
Description: as for outcome 12
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: Analysis was performed on AT analysis set which included all participants who received at least 1 dose of eliglustat during LIP.
Measure: Number; unit: participants
Arm/Group | LIP: Eliglustat
Number analyzed (Participants) | 170
participants
  MS,Unrestricted: Baseline (n=163) | 146
  MS,Unrestricted: Week 26 (n=161) | 153
  MS,Unrestricted: Week 52 (n=72) | 70
  MS,Unrestricted: Week 78 (n= 41) | 39
  MS, Walks With Difficulty: Baseline (n=163) | 12
  MS, Walks With Difficulty: Week 26 (n=161) | 6
  MS, Walks With Difficulty: Week 52 (n=72) | 1
  MS, Walks With Difficulty: Week 78 (n=41) | 2
  MS, Walks With Orthopedic Aid: Baseline (n=163) | 3
  MS, Walks With Orthopedic Aid: Week 26 (n=161) | 1
  MS, Walks With Orthopedic Aid: Week 52 (n=72) | 0
  MS, Walks With Orthopedic Aid: Week 78 (n=41) | 0
  MS, Required wheelchair: Baseline (n=163) | 2
  MS, Required wheelchair: Week 26 (n=161) | 1
  MS, Required wheelchair: Week 52 (n=72) | 1
  MS, Required wheelchair: Week 78 (n=41) | 0
  MS, Bedridden: Baseline (n=163) | 0
  MS, Bedridden: Week 26 (n=161) | 0
  MS, Bedridden: Week 52 (n=72) | 0
  MS, Bedridden: Week 78 (n=41) | 0

24. Secondary Outcome: LIP: Number of Participants With Bone Crises Assessment at Baseline, Weeks 26, 52 and 78
Description: Bone crises was assessed as a part of Gaucher disease assessment in participants. Acute, excruciating episodic bone pain is characteristic of Gaucher bone crises, which typically causes debilitation lasting several days or longer and requires treatment with immobilization, hydration, and opioid analgesics. Participants were categorized as 0= no bone crisis, 1= 1 bone crisis, 2= 2 bone crises, 6= 6 bone crises, and 24= 24 bone crises during the assessment period. In this outcome, number of participants with different bone crises levels at specified time points were reported.
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | LIP: Eliglustat
Number analyzed (Participants) | 170
participants
  Bone Crisis (0): Baseline (n=162) | 151
  Bone Crisis (0): Week 26 (n=162) | 159
  Bone Crisis (0): Week 52 (n=72) | 72
  Bone Crisis (0): Week 78 (n=41) | 41
  Bone Crisis (1): Baseline (n=162) | 8
  Bone Crisis (1): Week 26 (n=162) | 3
  Bone Crisis (1): Week 52 (n=72) | 0
  Bone Crisis (1): Week 78 (n=41) | 0
  Bone Crisis (2): Baseline (n=162) | 1
  Bone Crisis (2): Week 26 (n=162) | 0
  Bone Crisis (2): Week 52 (n=72) | 0
  Bone Crisis (2): Week 78 (n=41) | 0
  Bone Crisis (6): Baseline (n=162) | 1
  Bone Crisis (6): Week 26 (n=162) | 0
  Bone Crisis (6): Week 52 (n=72) | 0
  Bone Crisis (6): Week 78 (n=41) | 0
  Bone Crisis (24): Baseline (n=162) | 1
  Bone Crisis (24): Week 26 (n=162) | 0
  Bone Crisis (24): Week 52 (n=72) | 0
  Bone Crisis (24): Week 78 (n=41) | 0

25. Secondary Outcome: LIP: Number of Participants With Bone Pain Levels During the Past 4 Weeks at Baseline, Weeks 26, 52 and 78
Description: Bone pain was assessed as a part of Gaucher disease assessment in participants. Participants were categorized as none (no bone pain), very mild bone pain, mild bone pain, moderate bone pain, severe bone pain and extreme bone pain. In this outcome, number of participants with different type of bone pain during the past 4 weeks at specified time points were reported.
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | LIP: Eliglustat
Number analyzed (Participants) | 170
participants
  None: Baseline (n=163) | 112
  None: Week 26 (n=161) | 125
  None: Week 52 (n=72) | 62
  None: Week 78 (n=41) | 39
  Very Mild: Baseline (n=163) | 17
  Very Mild: Week 26 (n=161) | 14
  Very Mild: Week 52 (n=72) | 4
  Very Mild: Week 78 (n=41) | 1
  Mild: Baseline (n=163) | 22
  Mild: Week 26 (n=161) | 10
  Mild: Week 52 (n=72) | 3
  Mild: Week 78 (n=41) | 0
  Moderate: Baseline (n=163) | 8
  Moderate: Week 26 (n=161) | 10
  Moderate: Week 52 (n=72) | 3
  Moderate: Week 78 (n=41) | 1
  Severe: Baseline (n=163) | 4
  Severe: Week 26 (n=161) | 2
  Severe: Week 52 (n=72) | 0
  Severe: Week 78 (n=41) | 0
  Extreme: Baseline (n=163) | 0
  Extreme: Week 26 (n=161) | 0
  Extreme: Week 52 (n=72) | 0
  Extreme: Week 78 (n=41) | 0

26. Secondary Outcome: LTTP: Percentage of Participants Who Maintained a Stable Bone Criterion ,Hemoglobin Level, Platelet Count, Liver Volume and Spleen Volume at 1 Year and 2 Years
Description: Participant were considered as stable if they met the following criteria: hemoglobin level did not decrease >1.5 g/dL from baseline for PAP, platelet count does not decrease >25% below Baseline for PAP, liver volume does not increase >20% above Baseline for PAP, spleen volume does not increase >25% above Baseline for PAP. Baseline for PAP was defined as last available assessment prior to randomization.
Time Frame: 1 Year, 2 Years
Population: Analysis was performed on intent to treat (ITT) population which included all participants who received at least 1 dose of eliglustat after randomization. Here 'n' signifies number of participants with available data at specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- LTTP: Eliglustat: All participants who entered PAP continued their blinded randomized treatment for first 4 weeks. Participants who at Week 52 of PAP maintained their therapeutic goals (defined as: no more than 2 bone crisis during PAP [with no more than 1 bone crisis during either first 6 months or later 6 months of PAP] and is free of other clinically symptomatic bone disease during PAP; hemoglobin level not decreased by >1.5 g/dL from Baseline for PAP [defined as last available assessment prior to randomization]; platelet count not decreased by >25% from Baseline for PAP; spleen volume not increased by 25% from Baseline for PAP; liver volume not increased by >20% from Baseline for PAP), continued into the LTTP and received their TDD of eliglustat (100 mg or 200 mg) QD till the end of the study. The participants who did not maintain all their therapeutic goals continued into the LTTP and received their TDD of eliglustat (100 mg or 200 mg) BID till the end of the study.
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
percentage of participants
  Bone Criterion Stable at 1 year (n=104) | 92.3 [85.4 to 96.6]
  Bone Criterion Stable at 2 years (n=32) | 84.4 [67.2 to 94.7]
  Hemoglobin Level Stable at 1 year (n=104) | 92.3 [85.4 to 96.6]
  Hemoglobin Level Stable at 2 years (n=32) | 81.3 [63.6 to 92.8]
  Platelet Count Stable at 1 year (n=104) | 93.3 [86.6 to 97.3]
  Platelet Count Stable at 2 years (n=32) | 84.4 [67.2 to 94.7]
  Liver Volume Stable at 1 year (n=103) | 93.2 [86.5 to 97.2]
  Liver Volume Stable at 2 years (n=31) | 83.9 [66.3 to 94.5]
  Spleen Volume Stable at 1 year (n=72) | 95.8 [88.3 to 99.1]
  Spleen Volume Stable at 2 years (n=20) | 95.0 [75.1 to 99.9]

27. Secondary Outcome: LTTP: Number of Participants With Mobility Status (MS) at Baseline, 1 Year and 2 Years
Description: as for outcome 12
Time Frame: Baseline, 1 year, and 2 years
Population: All participants who received at least one dose of eliglustat during the LTTP.
Measure: Number; unit: participants
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
participants
  MS, Unrestricted: Baseline (n=120) | 111
  MS, Unrestricted: 1 year (n=104) | 97
  MS, Unrestricted: 2 years (n=32) | 28
  MS, Walks with Difficulty: Baseline (n=120) | 7
  MS, Walks with Difficulty: 1 year (n=104) | 4
  Ms, Walks with Difficulty: 2 years (n=32) | 2
  MS, Walks with Orthopedic Aid: Baseline (n=120) | 0
  MS, Walks with Orthopedic Aid: 1 year (n=104) | 1
  MS, Walks with Orthopedic Aid: 2 years (n=32) | 0
  MS, Required Wheelchair: Baseline (n=120) | 2
  MS, Required Wheelchair: 1 year (n=104) | 2
  MS, Required Wheelchair: 2 years (n=32) | 2
  MS, Bedridden: Baseline (n=120) | 0
  MS, Bedridden: 1 year (n=104) | 0
  MS, Bedridden: 2 years (n=32) | 0

28. Secondary Outcome: LTTP: Number of Participants With Bone Crises Assessment at Baseline, 1 Year and 2 Years
Description: Bone crises was assessed as a part of Gaucher disease assessment in participants. Acute, excruciating episodic bone pain is characteristic of Gaucher bone crises, which typically causes debilitation lasting several days or longer and requires treatment with immobilization, hydration, and opioid analgesics. Participants were categorized as 0= no bone crises, 1= 1 bone crisis during the assessment period. In this outcome, number of participants with different bone crises levels at specified time points were reported.
Time Frame: Baseline, 1 year and 2 years
Population: All participants who received at least one dose of eliglustat during the LTTP.
Measure: Number; unit: participants
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
participants
  Bone Crisis (0): Baseline (n=120) | 119
  Bone Crisis (0): 1 year (n=104) | 104
  Bone Crisis (0): 2 years (n=32) | 32
  Bone Crisis (1): Baseline (n=120) | 1
  Bone Crisis (1): 1 year (n=104) | 0
  Bone Crisis (1): 2 years (n=32) | 0

29. Secondary Outcome: LTTP: Number of Participants With Bone Pain Levels During the Past 4 Weeks at Baseline, 1 Year, and 2 Years
Description: Bone pain was assessed as a part of Gaucher disease assessment in participants. Participants were categorized as none (no bone pain), very mild bone pain, mild bone pain, moderate bone pain, severe bone pain and extreme bone pain. In this outcome, number of participants with different level of bone pain during the past 4 weeks at specified time points were reported.
Time Frame: Baseline, 1 year and 2 years
Population: All participants who received at least one dose of eliglustat during the LTTP.
Measure: Number; unit: participants
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
participants
  None: Baseline (n=120) | 91
  None: 1 year (n=104) | 83
  None: 2 years (n=32) | 32
  Very Mild: Baseline (n=120) | 12
  Very Mild: 1 year (n=104) | 9
  Very Mild: 2 years (n=32) | 0
  Mild: Baseline (n=120) | 8
  Mild: 1 year (n=104) | 10
  Mild: 2 years (n=32) | 0
  Moderate: Baseline (n=120) | 7
  Moderate: 1 year (n=104) | 1
  Moderate: 2 years (n=32) | 0
  Severe: Baseline (n=120) | 2
  Severe: 1 year (n=104) | 0
  Severe: 2 years (n=32) | 0
  Extreme: Baseline (n=120) | 0
  Extreme: 1 year (n=104) | 1
  Extreme: 2 years (n=32) | 0

30. Secondary Outcome: LTTP: Bone Mineral Density (BMD) at Baseline, 1 Year, and 2 Years
Description: BMD measurements of the spine and bilateral femur were acquired by DXA scan.
Time Frame: Baseline, 1 year, and 2 years
Population: All participants who received at least one dose of eliglustat during the LTTP.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
g/cm^2
  Lumbar Spine: Baseline (n=113) | 1.087 (0.182)
  Lumbar Spine: 1 year (n=101) | 1.083 (0.183)
  Lumbar Spine: 2 years (n=26) | 1.082 (0.190)
  Left Femur: Baseline (n=107) | 0.986 (0.205)
  Left Femur: 1 year (n=95) | 0.994 (0.226)
  Left Femur: 2 years (n=22) | 0.950 (0.220)
  Right Femur: Baseline (n=103) | 0.983 (0.201)
  Right Femur: 1 year (n=91) | 0.979 (0.202)
  Right Femur: 2 years (n=21) | 0.908 (0.131)

31. Secondary Outcome: LTTP: Total T-Scores for BMD at Baseline, 1 Year, and 2 Years
Description: as for outcome 10
Time Frame: Baseline, 1 year, and 2 years
Population: All participants who received at least one dose of eliglustat during the LTTP.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
T-score
  Lumbar Spine T-Score: Baseline (n=110) | -0.674 (1.383)
  Lumbar Spine T-Score: 1 year (n=98) | -0.718 (1.394)
  Lumbar Spine T-Score: 2 years (n=26) | -0.750 (1.370)
  Left Femur T-Score: Baseline (n=103) | -0.421 (1.377)
  Left Femur T-Score: 1 year (n=91) | -0.382 (1.551)
  Left Femur T-Score: 2 years (n=22) | -0.682 (1.532)
  Right Femur T-Score: Baseline (n=99) | -0.461 (1.360)
  Right Femur T-Score: 1 year (n=87) | -0.500 (1.381)
  Right Femur T-Score: 2 years (n=21) | -1.005 (0.931)

32. Secondary Outcome: LTTP: Total Z-scores for BMD at Baseline, 1 Year, and 2 Years
Description: as for outcome 11
Time Frame: Baseline, 1 year, and 2 years
Population: All participants who received at least one dose of eliglustat during the LTTP.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
Z-score
  Lumbar Spine Z-Score: Baseline (n=113) | -0.460 (1.376)
  Lumbar Spine Z-Score: 1 year (n=101) | -0.512 (1.368)
  Lumbar Spine Z-Score: 2 years (n=26) | -0.385 (1.316)
  Left Femur Z-Score: Baseline (n=107) | -0.164 (1.277)
  Left Femur Z-Score: 1 year (n=95) | -0.132 (1.459)
  Left Femur Z-Score: 2 years (n=22) | -0.264 (1.525)
  Right Femur Z-Score: Baseline (n=103) | -0.214 (1.227)
  Right Femur Z-Score: 1 year (n=91) | -0.262 (1.270)
  Right Femur Z-Score: 2 years (n=21) | -0.605 (0.957)

33. Secondary Outcome: LTTP: Total Bone Marrow Burden Score (BMB) at Baseline, 1 Year, and 2 Years
Description: BMB Score was measured using MRI, range from 0 (no abnormalities) to 8 points (severe disease) for the lumbar spine and from 0 (no abnormalities) to 8 points (severe disease) for the femurs. The total score was calculated as the sum of scores for femur and lumbar spine regions which ranged from 0 (no abnormalities) -16 (severe disease) points. A higher BMB score signified more severe bone marrow involvement.
Time Frame: Baseline, 1 year, and 2 years
Population: All participants who received at least one dose of eliglustat during the LTTP.
Measure: Mean (Standard Deviation); unit: BMB Score
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
BMB Score
  BMB Score: Baseline (n=115) | 8.164 (2.646)
  BMB Score: 1 year (n=26) | 7.853 (2.497)
  BMB Score: 2 years (n=17) | 8.059 (1.918)

34. Secondary Outcome: LTTP: Mean Biomarker (Chitotriosidase) Value at Baseline, 1 Year, and 2 Years
Description: Chitotriosidase biomarker was assayed from plasma.
Time Frame: Baseline, 1 year, and 2 years
Population: All participants who received at least one dose of eliglustat during the LTTP.
Measure: Mean (Standard Deviation); unit: nmol/hr/mL
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
nmol/hr/mL
  Chitotriosidase: Baseline (n=118) | 1188.983 (1857.521)
  Chitotriosidase: 1 year (n=97)) | 1221.753 (2072.446)
  Chitotriosidase: 2 years (n=31) | 598.161 (1463.603)

35. Secondary Outcome: LTTP: Mean Biomarker (GL-1 on DBS) Value at Baseline, 1 Year, and 2 Years
Description: GL-1 on DBS biomarker was assayed from dried blood spot.
Time Frame: Baseline, 1 year, and 2 years
Population: All participants who received at least one dose of eliglustat during the LTTP.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
mcg/mL
  GL-1 on DBS: Baseline (n=114) | 2.725 (1.350)
  GL-1 on DBS: 1 year (n=98) | 2.500 (1.031)
  GL-1 on DBS: 2 years (n=29) | 2.238 (0.658)

36. Secondary Outcome: LTTP: Mean Biomarker (MIP1-beta) Value at Baseline, 1 Year, and 2 Years
Description: MIP1-beta biomarker was assayed from plasma.
Time Frame: Baseline, 1 year, and 2 years
Population: All participants who received at least one dose of eliglustat during the LTTP.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LTTP: Eliglustat
Number analyzed (Participants) | 121
pg/mL
  MIP-1beta: Baseline (n=114) | 97.857 (125.857)
  MIP-1beta: 1 year (n=94) | 90.398 (90.549)
  MIP-1beta: 2 years (n=31) | 68.445 (64.774)

ADVERSE EVENTS:
Description: Adverse events data was planned to be reported for overall population.
Groups:
- Eliglustat: All participants who received eliglustat at the TDD of 100 mg or 200 mg in the LIP, PAP, LTTP or ETP.
Arm/Group | Eliglustat
Serious Adverse Events (participants affected / at risk) | 40/170
Other Adverse Events (participants affected / at risk) | 144/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eliglustat (N=170)
Angina pectoris (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Device dislocation (General disorders) | 1
Disuse syndrome (General disorders) | 1
Hernia (General disorders) | 1
Impaired healing (General disorders) | 1
Medical device pain (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Acute hepatitis B (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Hepatitis A (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 2
Ischaemic stroke (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Conversion disorder (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eliglustat (N=170)
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Palpitations (Cardiac disorders) | 11
Abdominal distension (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 15
Abdominal pain upper (Gastrointestinal disorders) | 26
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 24
Dyspepsia (Gastrointestinal disorders) | 19
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 14
Fatigue (General disorders) | 17
Pyrexia (General disorders) | 16
Hepatomegaly (Hepatobiliary disorders) | 9
Gastroenteritis (Infections and infestations) | 15
Influenza (Infections and infestations) | 23
Nasopharyngitis (Infections and infestations) | 52
Upper respiratory tract infection (Infections and infestations) | 22
Urinary tract infection (Infections and infestations) | 14
Viral infection (Infections and infestations) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 30
Back pain (Musculoskeletal and connective tissue disorders) | 29
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24
Dizziness (Nervous system disorders) | 28
Headache (Nervous system disorders) | 37
Depression (Psychiatric disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18
Hypertension (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.